CLINICAL TRIAL: NCT00222417
Title: Audiometric Parameters in Conductive Hearing Loss and Middle Ear Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: SFP-177-04/721170
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Otosclerosis; Tympanic Membrane Perforation
MeSH Terms: conditions — Otosclerosis; Tympanic Membrane Perforation | interventions — Myringoplasty; Stapes Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Myringoplasty: Patients subject to myringoplasty for tympanic membrane perforations.
  Interventions: Procedure: myringoplasty
- Otosclerosis: Patients subject to stapes surgery
  Interventions: Procedure: Stapes surgery

INTERVENTIONS:
Procedure: myringoplasty — Myringoplasty is an operative procedure to close tympanic membrane perforations.
  Groups: Myringoplasty
Procedure: Stapes surgery — Operative procedure aimed to replace non-functioning stapes with a synthetic prosthesis
  Groups: Otosclerosis

SUMMARY:
We study audiometric parameters including Transient Otoacoustic emissions, pure-tone audiometry for air- and bone-conduction, and spondaic speech recognition thresholds for air- and bone conduction in a pre- and postoperative situation in patients due for surgery for tympanic membrane perforations and otosclerosis. The hypotheses are that the precision of the preoperative assessment may be increased, and our knowledge about the effect on the inner ear by middle ear surgery may be increased.

DETAILED DESCRIPTION:
Consecutive patients 12 years or older due for myringoplasty or stapes surgery at the ENT-department, University hospital of Tromsø, in an approximate time span of one year, have been studied with the following audiometric investigations at the preoperative admission, 2, 6 and 12 months postoperatively: Transient otoacoustic emissions, pure-tone audiometry for air- and bone-conduction, speech audiometry using spondaic recognition for air and bone-conduction. Results will be statistically analysed using the Statistical Package for the Social Sciences, with the unoperated ear (paired organ) serving as controls. The goal is to look at alternative methods for analysing the patients' preoperative hearing in order to increase the precision of clinical decision-making. The secondary goal is to elucidate the effects of middle ear surgery on the inner ear.

ELIGIBILITY:
Inclusion Criteria:

* Tympanic membrane perforation without chronic secretion or cholesteatoma
* Suspected otosclerosis

Exclusion Criteria:

* Below 12 years of age
* Patient not consenting to study
* Perioperative findings suggesting chronic otitis or cholesteatoma
* Patients not fluent in Norwegian or unable to cooperate in audiometry

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sample of patients scheduled for middle ear surgery at the University Hospital North Norway in Tromsø.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2002-09; Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative hearing threshold level | 1 year
  Pure tone audiometry, speech audiometry, otoacoustic emissions

CONTACTS AND LOCATIONS:
Overall Officials: Niels C Stenklev, MD, PhD, Principal Investigator — ENT-department, University of Tromsø, 9038 Tromsø, Norway
Locations (1):
- ENT-department, University Hospital of Tromsø, Tromsø, Troms, Norway